CLINICAL TRIAL: NCT04529824
Title: Glucose Risk Assessment in Employer Populations
Status: Completed | Type: Observational
Sponsor: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PTL-903595
Record Dates: First submitted 2020-08-21; First posted 2020-08-28 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2022-03

CONDITIONS: Diabetes; Pre-diabetes; Glucose Intolerance
Keywords: continuous glucose monitoring; CGM
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance | interventions — Continuous Glucose Monitoring; Drug Delivery Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Dexcom G6 Continuous Glucose Monitor (CGM) System — Participants wear a blinded Dexcom G6 CGM and a Fitbit Charge 3 activity tracker for 10 days.
  Other Names: Fitbit Charge 3 Activity Tracker

SUMMARY:
This is an observational study to understand the glucose characteristics of the general population (normal glucose, pre-diabetes, and diabetes). Glucose risk will be measured with laboratory HbA1c and continuous glucose monitor (CGM) derived metrics. Physical activity will also be measured using a Fitbit activity tracker. The study will inform future programs that use CGM and activity tracking to identify people at risk for diabetes in the population.

DETAILED DESCRIPTION:
This is a prospective, single-center, observational study that will enroll a maximum of 550 subjects. All potential study subjects will be current or former employees or dependents eligible to enroll for Employer's group health plan and will demonstrate interest in response to recruitment materials placed in the near site clinic and/or the surrounding community. Participation interest will be demonstrated by calling the study number. Potential subjects will then undergo a screening call performed by study staff and, if still interested and likely eligible will be scheduled for Visit 1 and potential Visit 2. If a potential subject is not interested in continuing they will be given the option to anonymously complete a survey as to why they declined participation.

All potential subjects at Visit 1 will be required to provide written or electronic informed consent to participate. Once informed consent is obtained, study staff will confirm if there is a recent A1C available . If subject has a confirmed diagnosis of diabetes or pre-diabetes and an A1C result within the last 8-weeks or does not have diabetes or pre-diabetes and has an A1C within the last 6-months no A1C will be drawn. If the subject does not have a recent A1C a POC A1C will be taken at Visit 2. Study staff or subject will deploy the CGM system at Visit 1. Study staff will verify that the CGM is successfully blinded and subject has been trained on wearing CGM before subject completes Visit 1.

Subjects will be offered to wear an optional activity tracker and if chosen will also be required to download the activity tracker mobile application onto their personal smartphone. Subjects will then be trained on how to synchronize and charge their study activity tracker. To complete Visit 1 activities subjects will be asked to complete up to three surveys regarding their health status, reason for participation, diabetes risk, and if they decline to wear the activity tracker and why. Subjects upon leaving Visit 1 will confirm their return Visit 2 and remuneration will be processed at this time.

During the 10-day wear period subjects will have access to study staff in-person at the clinic and have Dexcom Technical Support available through a dedicated phone line Monday through Friday.

At Visit 2, study staff will assist subjects with removing the CGM and if wearing an activity tracker will also have it removed. Study staff will confirm the activity tracker has been synced with the subject's mobile application before deletion from the smartphone. Study staff will collect and record adverse events, serious adverse events, or unanticipated problems. Subjects will be asked to complete a user experience survey and have their mailing address confirmed for delivery of the final summary report and completion survey. A POC A1C will be obtained (unless a recent A1C and shared with subjects). Unless previously diagnosed with diabetes, subjects will be classified as normal glucose levels, prediabetes or diabetes based on their overall data. Subjects who are newly diagnosed with diabetes (POC A1C ≥ 6.5%) may be referred to their primary care physician. Remuneration will be processed at this time. Safety data will not be obtained for any subject after Visit 2 unless an ongoing AE is considered not resolved or ongoing and not stable.

Approximately 5 days after Visit 2, study staff will mail a final summary report of CGM and activity metrics along with a user experience survey together with a pre-addressed return envelope. The survey will provide the option for subjects to be called for follow-up interview by a study research staff trained in user-experience research for an interview about their experience. In addition, a subject data summary report may be provided to their primary care physician and/or endocrinologist. A majority of the subjects will be considered exited from the study after the interview or the interview was declined, and/or the user experience survey has been received. A select group of subjects (up to 50) will receive a new version of the data summary report based on the feedback collected from the initial group of completed data summary report surveys. Trained research staff will follow-up and discuss the changes with these subject.

36 months of retrospective and 24 months ± 1 month of prospective concurrent medical claims and cost data will be collected for each subject after the subject has been exited from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Current or former employee or dependent eligible to enroll in Employer's group health plan
2. Aged 18 years or older
3. Reads, speaks and understands English
4. Women of reproductive potential using one of the following highly effective modes of contraception: implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence or vasectomized partner.
5. Willing to comply with all study procedures (including CGM wear) and be available for the duration of the 10 day study
6. If a subject consents to optional wear of an activity tracker, the subject must:

   1. own a smartphone compatible with the Fitbit mobile application
   2. be willing to download the application on their smartphone
   3. be willing to use their assigned research account to sync data
   4. be willing to charge and sync data as directed during the 10 day wear

Exclusion Criteria:

1. Currently using continuous glucose monitoring
2. An intellectual or learning disability, or unstable mental state, that could limit ability to obtain written or electronic informed consent and/or adhere to the study protocol
3. Medical condition that precludes participation, including the following contraindications to CGM wear:

   1. Pregnant or planning to become pregnant
   2. Critically ill
4. Planned medical interventions that are listed as contraindications to CGM wear, including

   1. CT or MRI scan within 4 days of CGM insertion
   2. Dialysis
   3. Surgery
   4. Diathermy
5. Known skin issues and/or allergic reactions to components of the study product(s) (ex. medical-grade adhesives)
6. Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study.
7. Participation in another drug or device clinical trial concluding within 30 days of the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential volunteers will be adults (≥18 years) either currently or formerly employed by Employer and eligible to enroll for their health plan or added as dependents to the health plan.
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Diabetes Status | Clinic Visit 2 (about 10 days from study enrollment)
  diabetes status will be determined by A1C record or clinically measured point-of-care A1C (no diabetes <5.7%, pre-diabetes 5.7% to 6.4%, and diabetes > or = to 6.5%).

SECONDARY OUTCOMES:
CGM-derived Time in Range (TIR) | 10-days
  Estimated normal glucose time in range (TIR) (70-180 mg/dL)
CGM-derived Time Above Range (TAR) | 10-days
  Estimated time in hyperglycemia (>180 mg/dL)
CGM-derived Time Below Range (TBR) | 10-days
  Estimated time in hypoglycemia (<70 mg/dL)
CGM-derived Glucose Variability | 10-days
  Coefficient of variation of glucose (standard deviation/mean)
Fitbit-derived daily steps | 10-days
  average steps per day
Fitbit-derived light activity | 10-days
  average daily hours of light physical activity
Fitbit-derived moderate to vigorous activity | 10-days
  average daily minutes of moderate to light physical activity
Fitbit-derived sedentary time | 10-days
  average daily hours of sedentary time (< 3 METS)

OTHER OUTCOMES:
Healthcare medical costs | prior 3-years to study and 3-years after study participation
  Average monthly medical costs determined from medical claims billing data. Diagnosis and procedure codes are used to determine healthcare utilization (e.g., hospital stays, emergency room visits), which are converted to estimated costs to determine patient medical costs.

CONTACTS AND LOCATIONS:
Overall Officials: David Price, MD, Study Chair — DexCom, Inc.; Jennifer Ksailbati, CCRP, Principal Investigator — MOORE Clinical Research, Inc.
Locations (1):
- Lakeland Clinic, Lakeland, Florida, United States

IPD SHARING:
Plan to Share IPD: No